CLINICAL TRIAL: NCT01366963
Title: Origins of Cognitive Dysfunction in Postural Tachycardia Syndrome (POTS)
Brief Title: Cognitive Dysfunction in Postural Tachycardia Syndrome
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Satish R. Raj, Assistant Professor of Medicine, Vanderbilt University
Other Study IDs: 101401
Record Dates: First submitted 2011-02-17; First posted 2011-06-06 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Postural Tachycardia Syndrome
Keywords: postural tachycardia syndrome; brain fog; cognitive dysfunction
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Mental Fatigue; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Controls / Healthy Volunteers: Age and gender matched individuals without postural orthostatic tachycardia syndrome
  Interventions: Behavioral: Seated Measurements; Behavioral: Standing Measurements; Behavioral: Self-Administered Surveys
- Patients with Postural Tachycardia Syndrome (POTS): Individuals with Postural Tachycardia Syndrome
  Interventions: Behavioral: Seated Measurements; Behavioral: Standing Measurements; Behavioral: Self-Administered Surveys

INTERVENTIONS:
Behavioral: Seated Measurements — The following measurements will take place in a seated position:
  Ruff 1 & 7 (visual search and attention processes) Trails A & B (Tests of scanning, mental flexibility and executive processes) Symbol Digit Modalities Test (SDMT)(attention and psychomotor speed) Stroop Test (naming response to certain stimuli) Verbal Fluency (COWA) Randt Wechsler Test of Adult Reading (WTAR)
Behavioral: Standing Measurements — The following will be measured in a standing position (at least 5 minutes)
  Orthostatic Vital Signs Randt Paired Words Subtest Digits Forward and Backward Alternate COWA test
Behavioral: Self-Administered Surveys — Center for Epidemiologic Studies Depression Scale (CES-D) Cognitive-Somatic Anxiety Questionnaire (CSAQ) Subjective Neurocognitive Inventory (SNI)

SUMMARY:
A common complaint among people with Postural Tachycardia Syndrome (POTS) is "brain fog" or difficulty concentrating. This is very poorly understood. To better understand this cognitive dysfunction, the investigators will test people with POTS and people without POTS using various neuropsychiatric instruments. The investigators hypothesis is that people with POTS will have greater abnormalities on neuropsychiatric testing than normal controls.

DETAILED DESCRIPTION:
Postural Tachycardia Syndrome (POTS) is a disorder that affects an estimated 500,000 people in the United States alone and is an important source of disability in young adults. It shows a strong predilection for females. POTS is a form of orthostatic intolerance characterized by an excessive increase in heart rate (>30 bpm) on assuming the upright position associated with orthostatic symptoms, but in the absence of orthostatic hypotension. Their symptoms of dizziness, nausea, tremor, chronic fatigue and exercise intolerance make even simple activities of daily living exhausting prospects.

Brain fog or cognitive dysfunction is a common and almost universal complaint among persons with POTS. There is a lack of pathophysiological understanding to this cognitive dysfunction and is also a major roadblock to the development of effective therapies for people with POTS.

The purpose of this study is to better define the cognitive dysfunction seen in patients with POTS. We will use a series of validated neuropsychological tools in order to characterize POTS cognitive dysfunction and compare this data to age and gender matched control subjects.

Specific Aims:

1. To assess whether POTS patients have more neuropsychological abnormalities than control subjects during seated assessments.
2. To assess whether POTS patients have more neuropsychological abnormalities than control subjects during assessments while standing.
3. To ascertain the phenomenology of any neuropsychological deficits distinguishing POTS patients from controls.

ELIGIBILITY:
Inclusion Criteria:

All

* Ages between 18-60 years
* Male and female subjects are eligible
* Able and willing to provide informed consent

POTS - additional inclusion criteria - Diagnosed with postural tachycardia syndrome by Vanderbilt Autonomic Dysfunction Center (increase in heart rate greater than or equal to 30 beats per minute with position change from supine to standing (10 minutes; chronic symptoms consistent with POTS that are worse when upright and get better with recumbence.)

Control subjects - additional inclusion criteria

* Gender matched to POTS patients
* Age-matched to POTS patients (+/- 5 years of a POTS patient)
* Grossly matched in intelligence to POTS patients

Exclusion Criteria:

ALL

* Inability to give or withdrawal of informed consent
* Pregnancy (determined by patient self report)
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol.

POTS - additional exclusion criteria

- Overt cause for postural tachycardia (such as acute dehydration)

Normal Controls - additional exclusion criteria

* Previously diagnosed with Axis I psychiatric disorder
* Previously diagnosed learning disorder
* Previously diagnosed attention deficit hyperactivity disorder (ADHD)
* Prior psychosis
* past or present substance abuse
* History of loss of consciousness
* History of seizures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients having been diagnosed with postural tachycardia syndrome and age & gender matched normal controls
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Standing Digits Backwards Test | In the standing position for approximately 15 minutes. This is a cross-sectional study with no follow-up.
  This is a continuous variable that will provide a measure of attention with orthostatic stress.

SECONDARY OUTCOMES:
Cognitive Domain Score (CDS) | At seated and standing. This is a cross-sectional study without follow-up. All assessments are performed on a single day.
  The CDS will consist of
  1: Seated memory (Randt Short Story subtes, Paired words subtes and Digits Forward) and standing memory (Randt short story, paired words and digits forward).
  2. Seated Complex Attention (Ruff, SDMT, Trails A, Randt, Digits Backward) and standing complex attention (Randt digits backward) 3. Executive functioning only while standing (Stroop, Trails) 4. Seated and standing verbal fluency (COWA).

CONTACTS AND LOCATIONS:
Overall Officials: Satish Raj, MD, MSCI, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Raj V, Haman KL, Raj SR, Byrne D, Blakely RD, Biaggioni I, Robertson D, Shelton RC. Psychiatric profile and attention deficits in postural tachycardia syndrome. J Neurol Neurosurg Psychiatry. 2009 Mar;80(3):339-44. doi: 10.1136/jnnp.2008.144360. Epub 2008 Oct 31. PMID 18977825
- [Background] Ruff RM, Niemann H, Allen CC, Farrow CE, Wylie T. The Ruff 2 and 7 Selective Attention Test: a neuropsychological application. Percept Mot Skills. 1992 Dec;75(3 Pt 2):1311-9. doi: 10.2466/pms.1992.75.3f.1311. PMID 1484803
- [Background] Messinis L, Kosmidis MH, Tsakona I, Georgiou V, Aretouli E, Papathanasopoulos P. Ruff 2 and 7 Selective Attention Test: normative data, discriminant validity and test-retest reliability in Greek adults. Arch Clin Neuropsychol. 2007 Aug;22(6):773-85. doi: 10.1016/j.acn.2007.06.005. Epub 2007 Jul 20. PMID 17640850
- [Background] Tombaugh TN. Trail Making Test A and B: normative data stratified by age and education. Arch Clin Neuropsychol. 2004 Mar;19(2):203-14. doi: 10.1016/S0887-6177(03)00039-8. PMID 15010086
- [Background] Ruff RM, Light RH, Parker SB, Levin HS. Benton Controlled Oral Word Association Test: reliability and updated norms. Arch Clin Neuropsychol. 1996;11(4):329-38. PMID 14588937
- [Background] Schwartz GE, Davidson RJ, Goleman DJ. Patterning of cognitive and somatic processes in the self-regulation of anxiety: effects of meditation versus exercise. Psychosom Med. 1978 Jun;40(4):321-8. doi: 10.1097/00006842-197806000-00004. PMID 356080
- [Background] Moritz S, Kuelz AK, Jacobsen D, Kloss M, Fricke S. Severity of subjective cognitive impairment in patients with obsessive-compulsive disorder and depression. J Anxiety Disord. 2006;20(4):427-43. doi: 10.1016/j.janxdis.2005.04.001. Epub 2005 Jun 1. PMID 15935611
- [Background] Lezak MD, Howieson DB, Oring DW, Annay HJ, Isher JS. Neuropsychological Assessment. New York:Oxford University Press;2004
- [Background] Smith A. Symbol Digit Modalitites Test.Los Angeles:Western Psychological Services; 1982.
- [Background] Wechsler D. The Wechsler Test of Adult Reading. San Antonio, Texas: PsychCorp;2001.
- [Background] Radloff LS. The CES-D Scale: A self-report depression scale for resarch in the general population. Applied Psychological Measurement 1077;1:385-401.
- [Background] Putzke JD, Williams MA, Daniel FJ, Bourge RC, Boll TJ. Self-report versus performance based activities of daily living capacity among heart transplanta candidates and their caregivers. Journal of Clinical Psychology in Medical Settings 2000;7:121-32.